CLINICAL TRIAL: NCT02458846
Title: The Efficacy of a Visual Screening Program to Reduce Later Amblyopia and Untreated Refractive Errors
Brief Title: Efficacy of Visual Screening in Ontario
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Agnes Wong, Senior Scientist; Neurosciences and Mental Health, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000045972
Record Dates: First submitted 2015-01-08; First posted 2015-06-01 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Screened Schools (Experimental): 25 schools. Screening involved: crowded HOTV acuity test, Preschool Randot Stereoacuity Test, and Plusoptix autorefractor. Referral criteria followed AAPOS guidelines for screening for amblyopia and amblyopia risk factors. Children who fail any one of the three tests (including uncooperative/unable children) will be given a referral letter, which includes an assigned appointment time for a comprehensive eye exam at school with a licensed optometrist. Any needed glasses will be dispensed at no cost to the parents. 6 months after the eye exam, we will follow up with a phone call to parents to offer any additional support (such as replacing broken/lost glasses)
  Interventions: Other: Crowded HOTV Acuity Test; Other: Preschool Randot Stereoacuity Test; Device: Plusoptix Autorefractor; Other: Comprehensive Eye Exam
- Care As Usual Schools (No Intervention): 25 schools were randomly allocated to the "care as usual" schools. No intervention was provided by the research team, however, children may have received optometry/ophthalmology care via regular referral channels (e.g., family physicians, teachers)

INTERVENTIONS:
Other: Crowded HOTV Acuity Test — This is one of the most sensitive tests of acuity for vision screening of young children. The child is asked to recognize a letter (H,O,T,V) that is surrounded by bars to induce the crowding effects typical of amblyopia. Children were tested monocularly and was required to achieve at least 20/32 in each eye to pass. Children already wearing glasses were tested with their glasses on.
  Arms: Screened Schools
Other: Preschool Randot Stereoacuity Test — This is a reliable screening test for stereo depth perception for young children. Children wear polarized stereoglasses and are asked to identify or match shapes that are "hiding in the snow", which cannot be perceived if the child has abnormal binocular vision. Children were required to achieve at least 60 arcseconds of disparity to pass. Children already wearing glasses were tested with their glasses worn under the stereo glasses.
  Arms: Screened Schools
Device: Plusoptix Autorefractor — Autorefractors are electronic devices that measure refractive errors by focusing a light onto the child's eyes and recording how their reflections from the retina return to the camera. The Plusoptix has been shown to have high sensitivity and specificity in previous research. AAPOS (2013) guidelines were used to determine the referral criteria.
  Arms: Screened Schools
Other: Comprehensive Eye Exam — Children who did not pass all three screening tests were referred for full cycloplegic optometry exams, with a parent/guardian present. Optometrists assessed visual history, monocular visual acuity (near & far), strabismus, binocular function, abnormalities of the anterior segment, and cycloplegic refraction. If the optometrist prescribed glasses, frames were chosen at the time of the exam and the glasses were dispensed either at school (with an optician) or at the optometrist's office.
  Arms: Screened Schools

SUMMARY:
Amblyopia (lazy eye), is the leading treatable cause of vision loss in childhood. Uncorrected refractive errors (ie farsightedness) can lead to difficulties in school. Unfortunately, many children do not receive vision screening until they have already developed irreversible vision problems. We will conduct a cluster randomized clinical trial in which schools, not individual children, are randomly allocated to receive a kindergarten visual screening program or to receive no intervention by the research team (i.e., "care as usual"). We will compare the prevalence of visual problems (and proportion of children with reading problems) when the children are in Grade 2, after allowing for at least one year of treatment.

DETAILED DESCRIPTION:
The proposed study is a single-masked cluster randomized clinical trial, with randomization and analyses occurring at the level of "schools" (i.e., we are not randomly assigning individuals to groups). To assess the efficacy of a visual screening program, we will compare visual outcomes in 25 schools randomly chosen to receive the program and 25 schools allocated to "care as usual" one year after screening. The screening tools are HOTV crowded acuity, Preschool Randot Stereoacuity Test, and Plusoptix Autorefractor. The outcome measures will assess later differences between schools receiving the visual screening program and control schools for prevalence of (1) visual and (2) reading problems. A lower prevalence of either or both problems in schools where the visual screening program was offered would provide evidence for the efficacy of vision screening. Primary outcome measure is the prevalence of amblyopia, reduced stereo vision, and untreated clinically significant refractive errors in "screened" versus "care as usual" schools. Secondary outcome measure is the proportion of children performing 1 standard deviation below average on reading scores in "screened" versus "care as usual" schools.

ELIGIBILITY:
Inclusion Criteria:

* Screening: children enrolled in senior kindergarten (age 5-6 years)
* Follow-up: children enrolled in Grade 2 (age 7-8 years)

Exclusion Criteria:

• None

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2597 (Actual)
Dates: Start 2014-09; Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of amblyopia | 16 months
  Prevalence of suspected amblyopia, defined as 2-or-greater line difference in acuity between eyes
Prevalence of refractive errors | 16 months
  Untreated clinically significant refractive errors defined by AAPOS (2013) guidelines
Prevalence of reduced stereo vision | 16 months
  Stereoacuity is often reduced in patients with some types of amblyopia, and will defined as worse than 30 arcsec

SECONDARY OUTCOMES:
Proportion of below-average readers Year 1 | 10 months
  Proportion of Grade 1 children reading 1 SD below average
Proportion of below-average readers Year 2 | 22 months
  Proportion of Grade 2 children reading 1 SD below average

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Wong, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02458846/Prot_SAP_000.pdf